CLINICAL TRIAL: NCT01440946
Title: An Open-label, Multicenter Evaluation of Safety, Pharmacokinetics and Efficacy of Recombinant Coagulation Factor IX Fc Fusion Protein, BIIB029, in the Prevention and Treatment of Bleeding Episodes in Pediatric Subjects With Hemophilia B
Brief Title: Study of Recombinant Coagulation Factor IX Fc Fusion Protein, BIIB029, in Previously Treated Pediatric Participants With Hemophilia B
Acronym: Kids B-LONG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9HB02PED; 2011-003076-36 (EudraCT Number)
Record Dates: First submitted 2011-09-16; First posted 2011-09-27 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-08

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — factor IX Fc fusion protein; Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rFIXFc Prophylaxis (Experimental): At Baseline and at Day 1, participants receive a single intravenous (IV) injection of prestudy FIX and rFIXFc, respectively, over 10 (±5) minutes at a dose of 50 IU/kg. Immediately after the last PK sampling, the first prophylactic dose of approximately 50 to 60 IU/kg will be administered in clinic as an IV injection.
  Dose could be increased or decreased in increments of 10 IU/kg; increases to a maximum of 100 IU/kg and frequency of administration to a maximum of twice weekly, were allowed as indicated.
  Interventions: Drug: rFIXFc; Drug: FIX

INTERVENTIONS:
Drug: rFIXFc — Vials of rFIXFc were combined as needed, based on the actual labeled potency to achieve the participant's calculated dose. Partial vial use was allowed, in order to achieve the calculated dose.
  Other Names: BIIB029; recombinant coagulation factor IX Fc fusion protein; Alprolix®
Drug: FIX — Vials of prestudy FIX (provided by the participants) were combined as needed, based on the nominal labeled potency (e.g., 250 IU, 500 IU, and 1000 IU), to achieve the participant's calculated dose.
  Other Names: Factor IX

SUMMARY:
The primary objective of the study is to evaluate the safety of Recombinant Human Coagulation Factor IX Fc Fusion Protein (rFIXFc) in previously treated pediatric subjects with hemophilia B. Secondary objectives of this study in this study population are as follows: to evaluate the efficacy of rFIXFc for prevention and treatment of bleeding episodes; to evaluate and assess the pharmacokinetics (PK) of rFIXFc; to evaluate rFIXFc consumption for prevention and treatment of bleeding episodes

DETAILED DESCRIPTION:
At the Baseline visit (28 ± 7 days prior to Day 1), participants receive a single IV injection of prestudy FIX over 10 (±5) minutes in the clinic under medical supervision at a dose of 50 IU/kg. A washout period with no FIX treatment is required prior to administration of prestudy FIX and prior to rFIXFc. A PK assessment is done with prestudy FIX and also done with rFIXFc on Day 1. After completing the PK assessments, participants begin weekly prophylactic treatment with rFIXFc for approximately 50 weeks, to obtain 50 EDs. One ED is defined as a 24-hour period in which a participant received 1 or more doses of rFIXFc, with the time of the first injection of rFIXFc defined as the start of the ED.

ELIGIBILITY:
Key Inclusion Criteria:

* Severe hemophilia B defined as ≤ 2 IU/dl (≤ 2%) endogenous FIX
* Male < 12 years and weight ≥ 13 kg
* History of at least 50 documented prior exposure days to FIX
* No history of, or currently detectable, inhibitor

Key Exclusion Criteria:

* Other coagulation disorders in addition to Hemophilia B
* History of anaphylaxis associated with any FIX or IV immunoglobulin administration

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (15):
- United States (7):
  - Research Site, Phoenix, Arizona
  - Research Site, Sacramento, California
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Indianapolis, Indiana
  - Research Site, East Lansing, Michigan
  - Research Site, Pittsburgh, Pennsylvania
- Australia (2):
  - Research Site, Parkville, Victoria
  - Research Site, Subiaco, Western Australia
- Research Site, Dublin, Ireland
- Research Site, Utrecht, Netherlands
- Research Site, Johannesburg, South Africa
- United Kingdom (3):
  - Research Site, Basingstoke
  - Research Site, Cambridge
  - Research Site, London

REFERENCES:
- [Derived] Shapiro AD, Kulkarni R, Ragni MV, Chambost H, Mahlangu J, Oldenburg J, Nolan B, Ozelo MC, Foster MC, Willemze A, Barnowski C, Jain N, Winding B, Dumont J, Lethagen S, Barnes C, Pasi KJ. Post hoc longitudinal assessment of the efficacy and safety of recombinant factor IX Fc fusion protein in hemophilia B. Blood Adv. 2023 Jul 11;7(13):3049-3057. doi: 10.1182/bloodadvances.2022009230. PMID 36848635
- [Derived] Fischer K, Kulkarni R, Nolan B, Mahlangu J, Rangarajan S, Gambino G, Diao L, Ramirez-Santiago A, Pierce GF, Allen G. Recombinant factor IX Fc fusion protein in children with haemophilia B (Kids B-LONG): results from a multicentre, non-randomised phase 3 study. Lancet Haematol. 2017 Feb;4(2):e75-e82. doi: 10.1016/S2352-3026(16)30193-4. PMID 28159192

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants < 6 Years Old: At Baseline and at Day 1, participants received a single intravenous (IV) injection of prestudy FIX and rFIXFc, respectively, over 10 (±5) minutes at a dose of 50 IU/kg. Immediately after the last pharmacokinetic (PK) sampling, the first prophylactic dose of approximately 50 to 60 IU/kg was administered in clinic as an IV injection.
  Dose could be increased or decreased in increments of 10 IU/kg; increases to a maximum of 100 IU/kg and frequency of administration to a maximum of twice weekly, were allowed as indicated.
- Participants 6 to < 12 Years Old: At Baseline and at Day 1, participants received a single IV injection of prestudy FIX and rFIXFc, respectively, over 10 (±5) minutes at a dose of 50 IU/kg. Immediately after the last PK sampling, the first prophylactic dose of approximately 50 to 60 IU/kg was administered in clinic as an IV injection.
  Dose could be increased or decreased in increments of 10 IU/kg; increases to a maximum of 100 IU/kg and frequency of administration to a maximum of twice weekly, were allowed as indicated.
Period: Overall Study
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants < 6 Years Old; Participants 6 to < 12 Years Old: At Baseline and at Day 1, participants received a single IV injection of prestudy FIX and rFIXFc, respectively, over 10 (±5) minutes at a dose of 50 IU/kg. Immediately after the last PK sampling, the first prophylactic dose of approximately 50 to 60 IU/kg was administered in clinic as an IV injection.
  Dose could be increased or decreased in increments of 10 IU/kg; increases to a maximum of 100 IU/kg and frequency of administration to a maximum of twice weekly, were allowed as indicated.
- Total: Total of all reporting groups
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.6 (0.99) | 8.3 (1.45) | 5.5 (3.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Factor IX (FIX) Inhibitor Development
Description: An inhibitor test result ≥ 0.6 Bethesda units (BU)/mL, confirmed on 2 separate samples drawn 2 to 4 weeks apart, was considered positive. Both tests were to be performed by the central laboratory using the Nijmegen-modified Bethesda Assay. Incidences were summarized for any positive inhibitor for participants with ≥ 50 exposure days (EDs) to rFIXFc. In addition, the incidence for all participants, regardless of their EDs to rFIXFc, was also summarized. An exact 95% CI for the proportion of participants with a confirmed inhibitor was calculated using the Clopper-Pearson exact method for a binomial proportion.
Time Frame: Up to 50 weeks +/- 7 days, or up to 50 EDs if reached prior to Week 50
Population: Safety Analysis Set: participants who received at least 1 dose of prestudy FIX, or at least 1 dose of rFIXFc; n=number of participants with given number of EDs who had a valid inhibitor test.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: All Participants
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old | Total
Number analyzed (Participants) | 15 | 15 | 30
percentage of participants
  Participants with ≥ 50 EDs; n=10, 13, 23 | 0 [0 to 30.85] | 0 [0 to 23.16] | 0 [0 to 14.25]
  All participants regardless of # of EDs;n=15,15,30 | 0 [0 to 21.8] | 0 [0 to 21.8] | 0 [0 to 11.57]

2. Secondary Outcome: Annualized Bleeding Rate
Description: Annualized bleeding rate = (number of bleeding episodes during the efficacy period / total number of days during the efficacy period)*365.25. The efficacy period begins with the first prophylactic dose of rFIXFc and ends with the last dose (for prophylaxis or a bleeding episode). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. A bleeding episode started from the first sign of bleeding and ended no more than 72 hours after the last treatment for the bleeding episode, within which any symptoms of bleeding at the same location or injections less than or equal to 72 hours apart were considered the same bleeding episode. Any injection to treat the bleeding episode taken more than 72 hours after the preceding one was considered the first injection to treat a new bleeding episode at the same location. Any bleeding at a different location was considered a separate bleeding episode, regardless of time from last injection.
Time Frame: Up to 50 weeks +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc; based on the number of participants whose efficacy period was of at least 1 day in duration.
Measure: Median (Inter-Quartile Range); unit: bleeding episodes per participant per yr
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 15 | 15
bleeding episodes per participant per yr | 1.09 [0.00 to 2.90] | 2.13 [0.00 to 4.17]

3. Secondary Outcome: Annualized Joint Bleeding Rate (Spontaneous)
Description: Annualized bleeding rate for spontaneous joint bleeding episode=(number of bleeding episodes meeting those criteria during the efficacy period/total number of days during the efficacy period)*365.25. Efficacy period begins with the first prophylactic dose of rFIXFc and ends with the last dose (for prophylaxis or a bleeding episode). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. A bleeding episode started from the first sign of bleeding and ended ≤ 72 hours after the last treatment for the bleeding episode, within which any symptoms of bleeding at the same location or injections ≤ 72 hours apart were considered the same bleeding episode. Any injection to treat the bleeding episode taken > 72 hours after the preceding 1 was considered the first injection to treat a new bleeding episode at the same location. Any bleeding at a different location was considered a separate bleeding episode, regardless of time from last injection.
Time Frame: Up to 50 weeks +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc; based on the number of participants whose efficacy period is of at least 1 day in duration.
Measure: Median (Inter-Quartile Range); unit: bleeding episodes per participant per yr
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 15 | 15
bleeding episodes per participant per yr | 0.00 [0.00 to 1.2] | 0.00 [0.00 to 2.2]

4. Secondary Outcome: Participant Assessment of Response to Injections to Treat a Bleeding Episode
Description: Participant's assessment of the response (provided by the caregiver) to the first rFIXFc injection for each bleeding episode. Percentages were based on the number of bleeding episodes for which a response was provided for the first injection, using the following 4-point scale: excellent=abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hours after the initial injection; good=definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after an injection, but possibly requiring more than one injection after 24 to 48 hours for complete resolution; moderate=probable or slight beneficial effect within 8 hours after the initial injection and requiring more than one injection; no response=no improvement, or condition worsened, within approximately 8 hours after the initial injection.
Time Frame: Up to 50 weeks +/- 7 days
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc and had ≥ 1 bleeding episode; based on the number of injections with an evaluation.
Measure: Number; unit: percent of 1st injections w/ a response
Units Other Than Participants: Injections
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 9 | 11
Number analyzed (Injections) | 19 | 34
percent of 1st injections w/ a response
  Excellent or Good | 89.5 | 88.2
  Excellent | 52.6 | 41.2
  Good | 36.8 | 47.1
  Moderate | 5.3 | 11.8
  No Response | 5.3 | 0

5. Secondary Outcome: Physician's Global Assessment of the Participant's Response to His rFIXFc Regimen
Description: Investigators assessed each participant's response to his rFIXFc regimen using a 4-point scale: excellent=bleeding episodes responded to ≤ the usual number of injections or ≤ the usual dose of rFIXFc or the rate of breakthrough bleeding during prophylaxis was ≤ that usually observed; effective=most bleeding episodes responded to the same number of injections and dose, but some required more injections or higher doses, or there was a minor increase in the rate of breakthrough bleeding; partially effective=bleeding episodes most often required more injections and/or higher doses than expected, or adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses; ineffective=routine failure to control hemostasis, or hemostatic control required additional agents. Percentages are based on the total number of responses; multiple responses per participant are counted.
Time Frame: Up to 50 weeks +/- 7 days
Population: Full Analysis Set: participants who received ≥ 1 dose of rFIXFc; based on the number of responses.
Measure: Number; unit: percentage of responses
Units Other Than Participants: responses
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 15 | 15
Number analyzed (responses) | 48 | 59
percentage of responses
  Excellent | 85.4 | 89.8
  Effective | 14.6 | 10.2
  Partially Effective | 0 | 0
  Ineffective | 0 | 0

6. Secondary Outcome: Annualized rFIXFc Consumption by Type of Injection
Description: Annualized consumption of rFIXFc for prevention of bleeding (prophylactic), treatment of bleeding, and other rFIXFc injections. Consumption is calculated for the efficacy period. The efficacy period began with the first prophylactic dose of rFIXFc and ended with the last dose (regardless of the reason for dosing). Surgery/rehabilitation and PK evaluation periods were not included in the efficacy period. Annualized consumption = (total IU/kg of study treatment received during the efficacy period / total number of days during the efficacy period)*365.25. Participants who did not have a particular injection type are counted as having zero injections for that type.
Time Frame: Up to 50 weeks +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc.
Measure: Mean (Standard Deviation); unit: IU/kg rFIXFc per year
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 15 | 15
IU/kg rFIXFc per year
  Prophylactic injections | 3041.5 (577.55) | 3185.6 (683.71)
  Injections for bleeding | 147.9 (209.89) | 293.8 (515.59)
  Other injections | 29.2 (48.93) | 16.9 (44.90)

7. Secondary Outcome: Number of Days From the Last Prophylaxis Injection to a Spontaneous Bleeding Episode
Description: The number of days from the last prophylaxis injection to the onset of a new spontaneous bleeding episode, analyzed across all evaluable bleeding episodes per participant and per episode, based on the efficacy period. Evaluable bleeding episodes are those for which both a date and time are available for both the onset of the bleeding episode and the previous prophylactic injection. The efficacy period begins with the first prophylactic dose of rFIXFc and ends with the last dose (for prophylaxis or a bleeding episode). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. For 'Per participant' values, the number of days from the last prophylactic injection to a spontaneous bleeding episode is averaged across all evaluable spontaneous bleeding episodes per participant.
Time Frame: Up to 50 weeks +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc; number of participants and number of episodes were determined for participants with at least 1 evaluable spontaneous bleeding episode.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Evaluable Spontaneous Bleeding Episodes
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 4 | 6
Number analyzed (Evaluable Spontaneous Bleeding Episodes) | 5 | 11
days
  Per spontaneous bleeding episode | 3.97 [0.71 to 4.27] | 5.55 [3.30 to 6.04]
  Per participant | 4.12 [2.33 to 5.30] | 5.52 [4.41 to 6.04]

8. Secondary Outcome: Number of Injections Required for Resolution of a Bleeding Episode
Description: The number of injections required to resolve a bleeding episode per participant and per episode, based on the efficacy period. The efficacy period begins with the first prophylactic dose of rFIXFc and ends with the last dose (for prophylaxis or a bleeding episode). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. All injections given from the initial sign of a bleeding episode, until the last date/time within the bleeding episode window are counted. The resolution of a bleeding episode is defined as no sign of bleeding following injection for the bleeding episode. For 'Per participant' values, the number of injections required to resolve each bleeding episode is averaged across all bleeding episodes per participant.
Time Frame: Up to 50 weeks +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc; number of participants and number of episodes were determined for participants with at least 1 evaluable bleeding episode.
Measure: Median (Inter-Quartile Range); unit: injections
Units Other Than Participants: Bleeding Episodes
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 9 | 11
Number analyzed (Bleeding Episodes) | 22 | 38
injections
  Per bleeding episode | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Per participant | 1.0 [1.0 to 1.2] | 1.0 [1.0 to 1.7]

9. Secondary Outcome: Total Dose Required for Resolution of a Bleeding Episode
Description: The total dose required to resolve a bleeding episode per participant and per episode, based on the efficacy period. The efficacy period begins with the first prophylactic dose of rFIXFc and ends with the last dose (for prophylaxis or a bleeding episode). Surgery/rehabilitation periods and PK evaluation periods are not included in the efficacy period. For 'Per bleeding episode' values, for each bleeding episode, the total dose is the sum of the doses (IU/kg) administered across all injections given to treat that bleeding episode. For 'Per participant' values, the total dose (IU/kg) used to resolve each bleeding episode is averaged across all bleeding episodes per participant.
Time Frame: Up to 50 weeks +/- 7 days (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc; number of participants and number of episodes were determined for participants who had complete information on the dose administered to treat a bleeding episode.
Measure: Median (Inter-Quartile Range); unit: IU/kg
Units Other Than Participants: Bleeding Episodes
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 9 | 11
Number analyzed (Bleeding Episodes) | 22 | 38
IU/kg
  Per bleeding episode | 65.37 [50.68 to 125.00] | 89.77 [50.92 to 140.86]
  Per participant | 70.22 [55.40 to 97.22] | 52.22 [27.03 to 161.06]

10. Secondary Outcome: Maximum Plasma Activity (Cmax; One-stage Activated Partial Thromboplastin Time [aPTT] Clotting Assay)
Description: Cmax: maximum plasma FIX activity during a dosing interval. The values for Cmax were adjusted to the nominal dose of 50 IU/kg. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: Baseline (28±7 days before Day 1) Prestudy FIX Dosing: predose; 30±5 min, 3 hrs±30 min, 10±2 hrs, 24±3 hrs, 48±4 hrs postdose. Day 1 rFIXFc Dosing: predose; 30±5 min, 3 hrs ±30 min, 10±2 hrs, 24±3 hrs, 72±7 hrs, 120±12 hrs, 168±16 hrs postdose.
Population: PK Analysis Set: all participants with adequate PK data, defined as complete and evaluable PK samples through 168 hours after rFIXFc dosing. Complete means the availability of the 168-hour sample and at least enough other samples to allow for all the PK parameters to be estimated.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
IU/dL | 29.78 [26.18 to 33.87] | 35.84 [30.56 to 42.03]

11. Secondary Outcome: Terminal Half Life (t1/2; One-stage aPTT Clotting Assay)
Description: t1/2: time required for the concentration of the drug to reach half of its original value in the body. Non-compartmental methods. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
hours | 66.49 [55.86 to 79.14] | 70.34 [60.95 to 81.17]

12. Secondary Outcome: Clearance (CL; One-stage aPTT Clotting Assay)
Description: CL: the measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time. Non-compartmental methods. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
mL/h/kg | 4.365 [3.901 to 4.885] | 3.505 [3.006 to 4.087]

13. Secondary Outcome: Volume of Distribution at Steady State (Vss; One-stage aPTT Clotting Assay)
Description: Vss: volume of distribution at steady state. Non-compartmental methods. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
mL/kg | 365.1 [316.2 to 421.6] | 289.0 [236.7 to 352.9]

14. Secondary Outcome: Dose Normalized Area Under the Curve (DNAUC; One-stage aPTT Clotting Assay)
Description: DNAUC: dose normalized area under the drug concentration-time curve (extent of unmetabolized drug in circulation). Non-compartmental methods. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
IU*h/dL per IU/kg | 22.71 [20.32 to 25.38] | 28.53 [24.47 to 33.27]

15. Secondary Outcome: Mean Residence Time (MRT; One-stage aPTT Clotting Assay)
Description: MRT: the average time for all the drug molecules to reside in the body. Non-compartmental methods. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
hours | 83.65 [71.76 to 97.51] | 82.46 [72.65 to 93.60]

16. Secondary Outcome: Incremental Recovery (IR; One-stage aPTT Clotting Assay)
Description: IR for FIX activity following rFIXFc dosing: IU/dL rise in plasma FIX per IU/kg drug administered. Non-compartmental methods. The 95% confidence interval on the geometric mean is based on the t-statistic back-transformed from the log scale.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Number analyzed (Participants) | 11 | 13
IU/dL per IU/kg | 0.5898 [0.5152 to 0.6752] | 0.7170 [0.6115 to 0.8407]

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs): from informed consent up to 21 days after last dose; AEs: from Baseline (28 ± 7 days prior to Day 1) up to 14 (+7) days after last dose.
Description: Length of rFIXFc dosing was up to 50 weeks ± 7 days. Serious and non-serious AEs that were treatment-emergent with respect to rFIXFc are presented for those subjects in the Safety Analysis Set who were treated with rFIXFc.
Arm/Group | Participants < 6 Years Old | Participants 6 to < 12 Years Old
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/15
Other Adverse Events (participants affected / at risk) | 12/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants < 6 Years Old (N=15) | Participants 6 to < 12 Years Old (N=15)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Device Occlusion (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants < 6 Years Old (N=15) | Participants 6 to < 12 Years Old (N=15)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dental Caries (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 0
Seasonal Allergy (Immune system disorders) | 1 | 1
Croup Infectious (Infections and infestations) | 2 | 0
Ear Infection (Infections and infestations) | 2 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1
Gastroenteritis Norovirus (Infections and infestations) | 0 | 2
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 6
Oral Bacterial Infection (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 4 | 0
Accidental Drug Intake By Child (Injury, poisoning and procedural complications) | 1 | 0
Bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Face Injury (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Head Injury (Injury, poisoning and procedural complications) | 1 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Lip Injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Food Intolerance (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Abnormal Behaviour (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.